CLINICAL TRIAL: NCT04024020
Title: Chronic Insomnia and CSF Markers of Dementia
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 829221
Record Dates: First submitted 2019-07-15; First posted 2019-07-18 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with insomnia: Men and women with chronic insomnia (>5 years duration)
  Interventions: Other: lumbar puncture
- Good sleepers: Men and women with a longstanding pattern of good sleep
  Interventions: Other: lumbar puncture

INTERVENTIONS:
Other: lumbar puncture — Subjects will have a lumbar puncture to collect cerebrospinal fluid collection

SUMMARY:
The longstanding view has been that insomnia, and other forms of sleep disturbance, emerge as a consequence of dementia and are the result of progressive neuronal damage. However, there is growing evidence that the direction of causation may go both ways, with sleep disturbance potentially increasing vulnerability to dementia. Longitudinal studies have found that sleep disturbance often precedes and increases risk for dementia by several years.The purpose of this study is to examine the relationship between chronic insomnia and dementia biomarkers and orexin levels found in cerebrospinal fluid (CSF). Fifteen adults age 30-50 with chronic insomnia and age- and gender-matched good sleepers will undergo overnight polysomnography and CSF sampling in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-50
* Men and women
* To be included in the insomnia group, subjects must meet the following DSM5 Diagnostic Criteria for insomnia disorder: dissatisfaction with sleep quantity or quality (difficulty initiating or maintaining sleep, or waking up too early) despite adequate opportunity for sleep; sleep disturbance causes clinical significant distress or impairment in functioning; present at least 3 times per week for at least 3 months; sleep disturbance is not better explained by a medical or psychiatric condition or based on the effects of a substance

Exclusion Criteria:

* Diagnosis or evidence of sleep disorders other than insomnia as determined by the screening questionnaires and clinical history
* Women who have been pregnant or lactating within the past six months
* Non-fluency in spoken or written English
* Current or past month shiftwork defined as working during the evening or night shift
* Current use of medications or OTC products that impact sleep
* Evidence of neurological abnormalities that could include the risks associated with lumbar puncture (e.g.papilledema, mass lesion, Chiari malformation).

Ages: 30 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Adults with chronic insomnia and matched good sleepers
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gehrman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individuals With Insomnia | Good Sleepers
Started | 15 | 15
Completed | 13 | 13
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individuals With Insomnia | Good Sleepers | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (9.1) | 43.2 (9.2) | 43.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 12 | 8 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — This scale provides a measure of overall severity of insomnia, with higher scores indicating more severe symptoms. Scores range from 0 to 28.
  units on a scale | 16.5 (4.3) | 3.6 (3.7) | 10.1 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: CSF Markers Related to Dementia
Description: CSF levels of the proteins Abeta40 and Abeta42
Time Frame: one morning
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Individuals With Insomnia | Good Sleepers
Number analyzed (Participants) | 13 | 13
picograms per milliliter
  Abeta40 | 4332.1 (1250.5) | 4824.0 (2336.0)
  Abeta42 | 393.2 (122.8) | 419.4 (201.8)

2. Secondary Outcome: CSF Levels of Orexin
Description: Orexin is a chemical in the brain related to sleep regulation
Time Frame: one morning
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Individuals With Insomnia | Good Sleepers
Number analyzed (Participants) | 13 | 13
picograms per milliliter | 215.5 (11.9) | 214.5 (28.2)

ADVERSE EVENTS:
Time Frame: up to 1 month
Arm/Group | Individuals With Insomnia | Good Sleepers
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Individuals With Insomnia (N=15) | Good Sleepers (N=15)
headache (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The participants in this study had relatively mild insomnia, so it is not known whether the same pattern would be found for more severe cases. The size of this study is also relatively small so larger studies are needed to have more conclusive results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT04024020/Prot_SAP_000.pdf